CLINICAL TRIAL: NCT06487624
Title: A Phase 1, Open-label, Multicenter, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of HCB301 in Subjects With Advanced Solid Tumors or Relapsed and Refractory cHL
Brief Title: An Engineered Sirpα Fused to Anti-Pd-L1 And Tgf-β Fusion Protein (HCB301) in Subjects With Selected Advanced Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: FBD Biologics Limited (Industry)
Collaborators: HanchorBio Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HCB301-101
Record Dates: First submitted 2024-06-24; First posted 2024-07-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor; Refractory Hodgkin Lymphoma
Keywords: Immunotherapy; CD47; PD-L1; TGF-beta; Tumor; Cancer
MeSH Terms: conditions — Hodgkin Disease; Camurati-Engelmann Syndrome; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Experimental: 0.3 mg/kg HCB301 (Experimental): 0.3 mg/kg HCB301 in subjects with advanced solid tumors or relapsed and refractory classical Hodgkin lymphomas.
  Interventions: Drug: HCB301
- Experimental: 0.6 mg/kg HCB301 (Experimental): 0.6 mg/kg HCB301 in subjects with advanced solid tumors or relapsed and refractory classical Hodgkin lymphomas.
  Interventions: Drug: HCB301
- Experimental: 1.2 mg/kg HCB301 (Experimental): 1.2 mg/kg HCB301 in subjects with advanced solid tumors or relapsed and refractory classical Hodgkin lymphomas.
  Interventions: Drug: HCB301
- Experimental: 2.4 mg/kg HCB301 (Experimental): 2.4 mg/kg HCB301 in subjects with advanced solid tumors or relapsed and refractory classical Hodgkin lymphomas.
  Interventions: Drug: HCB301
- Experimental: 4.8 mg/kg HCB301 (Experimental): 4.8 mg/kg HCB301 in subjects with advanced solid tumors or relapsed and refractory classical Hodgkin lymphomas.
  Interventions: Drug: HCB301
- Experimental: 9.6 mg/kg HCB301 (Experimental): 9.6 mg/kg HCB301 in subjects with advanced solid tumors or relapsed and refractory classical Hodgkin lymphomas.
  Interventions: Drug: HCB301
- Experimental: 15.0 mg/kg HCB301 (Experimental): 15.0 mg/kg HCB301 in subjects with advanced solid tumors or relapsed and refractory classical Hodgkin lymphomas.
  Interventions: Drug: HCB301

INTERVENTIONS:
Drug: HCB301 — HCB301 administered via. intravenous (IV) infusion.
  Other Names: 2023-3979 Solid Tumors

SUMMARY:
The purpose of this study is to find out whether IV injection of HCB301 is an effective treatment for different types of advanced solid tumors and relapsed and refractory classical Hodgkin lymphomas and what side effects (unwanted effects) may occur in subjects aged 18 years old and above.

DETAILED DESCRIPTION:
This is a phase 1, open-label, multicenter, dose-escalation study. This study is to evaluate the safety, tolerability, pharmacokinetics (PK), preliminary efficacy, and identification of maximum tolerated dose (MTD) of HCB301 intravenous injection in adults with advanced solid tumors or relapsed and refractory classical Hodgkin lymphomas.

Eligible subjects must have failed standard therapies, been intolerable, or been considered medically inappropriate by the investigator. Subjects will be treated until unacceptable AEs, radiographic or clinical documented disease progression, withdrawal of consent, loss to follow-up, death, or termination of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and be willing to sign the ICF.
2. Male and female subjects of ≥18 years of age.
3. Histologically/cytologically confirmed, locally advanced solid tumor:

   subjects confirmed advanced solid tumors who have relapsed or refractory and should have no options for standard or approved therapies known to potentially confer clinical benefit or classical Hodgkin lymphoma, relapsed or refractory to at least 2 prior lines of systemic therapy.
4. For subjects with advanced solid tumors - must have at least 1 measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 at baseline.
5. For subjects with classical Hodgkin lymphoma - must have classical Hodgkin lymphoma that is measurable or assessable for response.
6. Must have ECOG performance status of 0 to 1 at Screening.
7. Able to provide tumor tissue samples.
8. Have a life expectancy of ≥12 weeks.

Exclusion Criteria:

1. With known history of hypersensitivity to any components of HCB301.
2. Known active or untreated CNS metastases and/or carcinomatous meningitis.
3. Have undergone a major surgery or radical radiotherapy within 28 days or palliative radiotherapy within 14 days or have used a radioactive drug within 56 days prior to the first dose of HCB301.
4. Clinically significant cardiovascular condition.
5. Any previous treatment-related toxicities which have not recovered to ≤ Grade 1 as evaluated by National Cancer Institute, Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 or baseline, except alopecia and anemia.
6. With known inherited or acquired bleeding disorder or bleeding diathesis. .
7. Have RBC transfusion within 4 weeks prior to Screening.
8. With a previously documented diagnosis of hemolytic anemia or Evans Syndrome in the last 3 months.
9. Any investigational or approved systemic cancer therapy administered within 21 days or 5 half-lives, whichever is shorter, before the first dose of the study drug.
10. Active use of vitamin K antagonist anticoagulant like warfarin. Use of low molecular weight heparin and factor Xa inhibitors will be permitted on case by case basis. There will be no restriction for daily aspirin ≤ 100 mg/QD.
11. Have used herbal medication within 14 days prior to the first dose of HCB301.
12. Have received any treatment targeting the SIRPα-CD47, PD-L1, or TGF-β pathway.
13. Have other malignancies requiring treatment within 2 years prior to the first dose of HCB301.
14. An investigational device used within 28 days prior to the first dose of HCB301.
15. Positive for hepatitis B, active hepatitis C infections, positive for HIV, or known active or latent tuberculosis.
16. Known to have a history of alcoholism or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Number/incidence and percentage of subjects with adverse events, including ADA. | 12 months
  To evaluate the safety and tolerability of HCB301.
Number of subjects with MTD and RDE of HCB301. | 12 months
  To determine the MTD and RDE.

SECONDARY OUTCOMES:
Overall Rate Response (ORR) | 12 months
  ORR is defined as the proportion of participants who have a partial response (PR) or critical response (CR).
Duration of Response (DoR) | 12 months
  DoR is defined as time from date of initial documentation of a response (PR or CR) to date of first documented evidence of progressive disease (PD).
Disease Control Rate (DCR) | 12 months
  DCR is defined as the proportion of participants who have a partial response (PR), critical response (CR), or disease stable (SD).
Progression-Free Survival (PFS) | 12 months
  Defined as the duration from the start of treatment until tumor progression or death of any cause.
Peak Plasma Concentration (Cmax) of HCB301 | 12 months
  Peak Plasma Concentration (Cmax) of HCB301 following single and repeated IV doses of HCB301 at different dose levels.
Area under the plasma concentration versus time curve (AUC) of HCB301 | 12 months
  Area under the plasma concentration versus time curve (AUC) of HCB301 following single and repeated IV doses of HCB301 at different dose levels.
Time to maximum drug concentration in plasma (Tmax) of HCB301 | 12 months
  Time to maximum drug concentration in plasma (Tmax) of HCB301 following single and repeated IV doses of HCB301 at different dose levels.
Terminal elimination half-life (t1/2) of HCB301 | 12 months
  Terminal elimination half-life (t1/2) of HCB301 following single and repeated IV doses of HCB301 at different dose levels.

OTHER OUTCOMES:
CD47 receptor occupancy on circulating red blood cells (RBCs) | 12 months
  CD47 receptor occupancy on circulating red blood cells (RBCs) will be measured as an indication of target engagement.
Concentration of potential PD biomarkers in participants will be assess. | 12 months
  Changes in CD47 receptor occupancy on circulating CD3+ T cells and TGFβ1, 2, 3 will be assessed after HCB301 treatment.
ctDNA detection | 12 months
  ctDNA detection in participants using next-generation sequencing (NGS ).

CONTACTS AND LOCATIONS:
Locations (6):
- Prisma Health-Upstate, Greenville, South Carolina, United States
- China (5):
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Provincial Cancer Hospital, Hangzhou
  - Xuzhou Central Hospital, Xuzhou
  - Yantai Yuhuangding Hospital, Yantai
  - Southern Medical University Zhujiang Hospital, Zhujiang